CLINICAL TRIAL: NCT02700880
Title: Prospective Registry of Patients With Ischemic Heart Failure Using the LifeVest Wearable Cardioverter Defibrillator (WEARIT-III)
Brief Title: LifeVest Wearable Cardioverter Defibrillator WEARIT-III Registry
Acronym: WEARIT-III
Status: Completed | Type: Observational
Sponsor: Zoll Medical Corporation (Industry)
Collaborators: University of Rochester (Other)
Responsible Party: Sponsor
Other Study IDs: WEARIT-III
Record Dates: First submitted 2016-02-25; First posted 2016-03-07 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Ischemic Heart Failure
Keywords: wearable cardioverter defibrillator; ischemic cardiomyopathy; new onset heart failure; sudden cardiac death
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Heart failure patients with LifeVest: Subjects with ischemic cardiomyopathy and heart failure (including NYHA II, III, IV and an ejection fraction ≤ 35%) who wear a medically prescribed ZOLL LifeVest Wearable Defibrillator
  Interventions: Device: LifeVest

INTERVENTIONS:
Device: LifeVest — LifeVest monitors patients for VT/VF, notifies the patient if VT/VF occurs, and instructs them to press response buttons. In unresponsive patients, LifeVest delivers defibrillation therapy.
  Other Names: Wearable Cardioverter Defibrillator WCD

SUMMARY:
The WEARIT-III registry enrolls subjects with ischemic cardiomyopathy and heart failure (including NYHA II, III, IV and an ejection fraction ≤ 35%) who wear a medically prescribed ZOLL LifeVest Wearable Defibrillator. The primary objective of the WEARIT-III Registry is to prospectively document the clinical course of high-risk cardiac patients with heart failure and ischemic cardiomyopathy prescribed with Wearable Cardioverter Defibrillator (WCD), such as left ventricular function recovery, arrhythmia, Implantable Cardioverter Defibrillator (ICD), Cardiac Resynchronization Therapy (CRT), Left Ventricular Assist Device (LVAD), heart transplantation, and to assess the benefit of WCD in heart failure patients with ischemic cardiomyopathy.

DETAILED DESCRIPTION:
STUDY PROCEDURE

U.S. patients prescribed a commercially available WCD (ZOLL LifeVest) will be approached by a letter from the sponsor which summarized the study purpose and procedure. Once a patient signs a consent form to participate the study, he or she will receive three questionnaire from University of Rochester, the coordination and data center for the WEARIT registry, at the time enrollment, at 3 month and 12 month follow-up, respectively. At 3 and 12-month follow-up, the physician of the patient will be contacted to provide information on arrhythmias, and interim events (ICD, CRT or LVAD implantation, heart failure episode, death), and to send us related hospital reports and echocardiogram reports to assess the improvement in left ventricular function.

STUDY DESIGN

WEARIT-III is a prospective observational patient registry. Optimal pharmacologic and/or implanted device therapy is anticipated, and the Registry physicians will not be involved in any medical care of the subjects, only collecting information on the standard care of these patients. In WEARIT-III we will also retrieve hospital records/echocardiogram reports of the subjects during follow-up using an authorization form signed by the study subjects and contact their physician to collect information on improvement of the left ventricular function whenever it is available.

DATA MANAGEMENT, DATA STORAGE

Once consented, device recordings and prescribing information will be obtained from the device provider. Data from the subject-completed questionnaire will also be obtained. Data will be entered into our web-based, password-protected clinical data-management system. That data will then be doubled-checked for accuracy by personnel working on the Registry. All study documents will be kept in a locked file room. All computers are password-protected and kept in a locked area.

DATA ANALYSIS

Routine patient clinical data as well as WCD data and clinical outcome during 1 year of follow-up will be recorded on all study patients and entered into a study-specific data- management system using our existing data management systems in the Heart Research Follow-up Program.

All analyses will be performed based on the primary and secondary objectives. Patient's clinical characteristics will be recorded and presented by descriptive statistics. Change in the clinical course will be recorded by descriptive statistics and compared to pre- WCD and post-WCD. Time-to-event analysis will be performed to assess the time until medication optimization. Clinical event will be presented as person-time rate and will be compared to previous WCD studies. Adverse events will be evaluated by raw counts and percentages. Compliance will be analyzed by mean and median of length of use and daily wear time.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of 18 years old or older;
2. Subjects who are recently diagnosed with heart failure of ischemic etiology (either revascularized or cannot be revascularized);
3. NYHA functional class II, III, or IVa (ambulatory);
4. Left ventricular ejection fraction ≤ 35%;
5. Subject wearing a prescribed ZOLL LifeVest WCD;
6. Subject agrees to enter the Registry after appropriate informed consent.

Exclusion Criteria:

1. Subjects who are unable or unwilling to cooperate with the study protocol;
2. Subjects who are not willing to participate;
3. Subjects who have acute ST-segment elevation myocardial infarction (STEMI) within 30 days before prescribed with WCD;
4. Subjects with cardiomyopathy from mixed etiology;
5. Subjects with active or previously explanted cardiac devices such as ICD, CRT or LVAD except for pacemaker;
6. Subjects with a life expectancy of less than a year, including end-stage heart failure, cancer and end-stage renal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In WEARIT-III, subjects with ischemic cardiomyopathy and heart failure (including NYHA II, III, IV and an ejection fraction ≤ 35%) who wear a medically prescribed ZOLL LifeVest Wearable Cardioverter Defibrillator (WCD) and agree to enter the Registry after appropriate informed consent will be enrolled.
  It is anticipated that approximately 1000 patients with ischemic cardiomyopathy and heart failure (≥18 years of age) will be enrolled in 2 years. No individuals shall be excluded from participation in the Registry based on race, ethnicity or gender.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Number of clinical events in heart failure patients with ischemic cardiomyopathy prescribed wearable cardioverter defibrillator (WCD) | 1 year
  The primary objective of the WEARIT-III Registry is to prospectively document the clinical course of high-risk cardiac patients with heart failure and ischemic cardiomyopathy prescribed with WCD, such as left ventricular function recovery, arrhythmia, implantable cardioverter defibrillator (ICD), cardiac resynchronization therapy (CRT), left ventricular assist device (LVAD), heart transplantation, and to assess the benefit of WCD in heart failure patients with ischemic cardiomyopathy.

SECONDARY OUTCOMES:
All-cause mortality | 1 year
  Evaluate the number of deaths and the cause of death in patients with ischemic cardiomyopathy and heart failure prescribed with WCD.
Number of inappropriate shocks | 1 year
  Evaluate the safety of WCD in patients with ischemic cardiomyopathy and heart failure measured by the frequency of inappropriate WCD shocks
WCD shock conversion success rate | 1 year
  Evaluate WCD shock efficacy measured by shock conversion success rate among WCD appropriate shocks
NYHA functional class | At enrollment, 3-month and 1-year follow-up
  Evaluate the NYHA functional class of heart failure patients with ischemic cardiomyopathy at enrollment, 3-month and 1-year after the initial prescription of the WCD in WEARIT-III

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Kutyifa, MD,PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No